CLINICAL TRIAL: NCT01733784
Title: Mechanisms of Pharyngeal Collapse in Sleep Apnea, Study D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012P000957D; 1R01HL102321-01A1 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-27 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Sleep Apnea
Keywords: Sleep Apnea; Pathophysiology
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Viscoelastic properties of the airway (Experimental)
  Interventions: Other: Induced central apneas

INTERVENTIONS:
Other: Induced central apneas

SUMMARY:
In obstructive sleep apnea (OSA), the upper airway recurrently closes during sleep. The mechanisms that lead to airway closure are not completely understood. Some studies have shown that there is progressive narrowing of the pharyngeal airway across breaths during expiration (Progressive Expiratory Narrowing, PEN) preceding an obstructive apnea. The investigators will assess the viscoelastic properties of the pharyngeal airway and its role in PEN.

DETAILED DESCRIPTION:
In obstructive sleep apnea, the upper airway recurrently closes during sleep. The mechanisms that lead to airway closure are not completely understood. Some studies have shown that there is progressive narrowing of the pharyngeal airway across breaths during expiration (Progressive Expiratory Narrowing, PEN) preceding an obstructive apnea.

The investigators will test how the viscoelastic properties of the airway influence PEN. To this end, the investigators will visualize the pharynx of sleep apnea patients using a thin endoscope and will induce central apneas during sleep. Pharyngeal cross-sectional area will be recorded during incremental changes in pharyngeal pressure during central apneas.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects or patients with OSA

Exclusion Criteria:

* Any unstable cardiac condition (other than well controlled hypertension) or pulmonary problems.
* Any medication known to influence breathing, sleep/arousal or muscle physiology
* Concurrent sleep disorders (insomnia, narcolepsy, central sleep apnea or parasomnia)
* Claustrophobia
* Inability to sleep supine
* Allergy to lidocaine or oxymetazoline hydrochloride
* For women: Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12-08 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Upper airway elasticity | 10 - 40 seconds
  The investigators will determine elasticity of the upper airway during induced central apneas by dividing the change in airway pressure by the change in airway cross-sectional area.
  The time frame for the outcome of this study is equal to the duration of the induced central sleep apnea (usually less than 40 seconds).

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States